CLINICAL TRIAL: NCT04984993
Title: A Multi-centre, Randomised, Open-label, Home Use, Parallel Group, Clinical Investigation of Topically-applied MED3000 Gel and Oral Tadalafil (5 mg) Tablets for the Treatment of Erectile Dysfunction (ED) Over a 24 Week Period
Brief Title: Clinical Investigation Using MED3000 Gel or Tadalafil Tablets in the Treatment of Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Futura Medical Developments Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM71
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2021-07

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to receive either MED3000 gel or tadalafil (5 mg) tablets after a 4 -6 week screening period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- MED3000 (Experimental): MED3000 gel formulation topically applied to the glans penis
  Interventions: Device: MED3000 (Male); Device: MED3000 (Female)
- Tadalafil (Experimental): Tadalafil (5 mg) tablets to be taken orally
  Interventions: Drug: Tadalafil 5mg (Male); Drug: Tadalafil 5mg (Female)

INTERVENTIONS:
Device: MED3000 (Male) — Gel formulation
  Arms: MED3000
Drug: Tadalafil 5mg (Male) — Tablets
  Arms: Tadalafil
Device: MED3000 (Female) — Gel formulation
  Arms: MED3000
Drug: Tadalafil 5mg (Female) — Tablets
  Arms: Tadalafil

SUMMARY:
An open-label investigation using MED3000 gel or tadalafil (5 mg) tablets in the treatment of erectile dysfunction in patients from 22 to 70 years of age. Each patients will be expected to participate for up to 30 weeks. Eligible patients will be randomised to receive either MED3000 gel or tadalafil (5 mg) tablets in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Male heterosexual patients aged 22-70 years.
* Confirmed clinical diagnosis of mild, moderate or severe ED for more than 3 months.
* Involved in a continuous heterosexual relationship with their partner for at least 6 months.

Exclusion Criteria:

* Any significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological or psychiatric disease.
* History of unstable medical or psychiatric condition or using any medication that, in the opinion of the Principal Investigator, is likely to affect the patient's ability to complete the investigation or precludes the patient's participation in the investigation.

Ages: 22 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients who have had erectile dysfunction for at least 3 months
Enrollment: 116 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Burnett, MD, Principal Investigator — Johns Hopkins University
Locations (18):
- Johns Hopkins University, Baltimore, Maryland, United States
- Bulgaria (5):
  - Medical Center "Asklepii"OOD, Dupnitsa
  - ЕТ "Аssoc. Prof. Stefan Popov - Individual Practice for Specialized Outhospital medical care for Neurology and Pscyhiatry", Plovdiv
  - UMHAT Plovdiv AD, Plovdiv
  - MHAT "Silistra"AD, Silistra
  - Medical Center "INTERMEDICA"ООD, Sofia
- Georgia (6):
  - LTD Health, Batumi
  - Jsc "Evex Clinics", Kutaisi
  - Rustavi N2 Medical Diagnostic Center, Rustavi
  - Clinic "GIDMEDI", Tbilisi
  - JSC "Evex clinics", Tbilisi
  - Raymann LLC, Tbilisi
- Poland (6):
  - The Mikolowska Medical Center, Katowice
  - Provita Sp. z o.o., Katowice
  - Medistica Osteomed, Krakow
  - PROVITA Specialised Gynecology and Sexology Practice, Lublin
  - Sexology and Pathology of Intercourse Clinic, Warsaw
  - Ryszard Smoliński's Medical Cabinet, Wroclaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first informed consent was on September 14, 2021 and the last study visit was on June 13, 2022.
Pre-assignment Details: Of 232 screened patients (males and females enrolled for eligibility assessment), 192 patients and their partners were randomised to treatment. Of the 40 patients and partners that failed screening, 36 did not satisfy inclusion criteria and 2 were excluded for other reasons.
Groups:
- MED3000: MED3000 gel formulation topically applied to the glans penis
  MED3000: Gel formulation
- Tadalafil: Tadalafil (5 mg) tablets to be taken orally
  Tadalafil 5mg: Tablets
Period: Overall Study
Arm/Group | MED3000 | Tadalafil
Started | 96 | 96
Received Treatment | 94 | 94
Completed | 82 | 92
Not Completed | 14 | 4
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Both patients moved to another country | 4 | 0

BASELINE CHARACTERISTICS:
Population: Regional enrolment details are combined for both the male participants and their female partners.
Groups:
- Total: Total of all reporting groups
Arm/Group | MED3000 | Tadalafil | Total
Number analyzed (Participants) | 96 | 96 | 192
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Data are presented separately for male participants and female partners.
  Years
    Male: number analyzed (Participants) | 48 | 48 | 96
    Male | 46.1 (13.5) | 41.5 (11.5) | 43.8 (12.7)
    Female: number analyzed (Participants) | 48 | 48 | 96
    Female | 43.3 (13.9) | 40.0 (11.5) | 41.6 (12.8)
Age, Continuous [Median (Full Range); unit: Years] — Population: Data are presented separately for male participants and female partners.
  Years
    Male: number analyzed (Participants) | 48 | 48 | 96
    Male | 44.5 [22 to 68] | 39.0 [23 to 68] | 40.5 [22 to 68]
    Female: number analyzed (Participants) | 48 | 48 | 96
    Female | 39.5 [20 to 69] | 38.0 [19 to 65] | 39.0 [19 to 69]
Age, Customized [Count of Participants; unit: Participants] — Population: Data are presented separately for male participants and female partners.
  Participants
    Male: number analyzed (Participants) | 48 | 48 | 96
    Male: 22-29 | 5 | 7 | 12
    Male: 30-39 | 16 | 18 | 34
    Male: 40-49 | 5 | 13 | 18
    Male: 50-59 | 10 | 5 | 15
    Male: 60-70 | 12 | 5 | 17
    Male: <22 | 0 | 0 | 0
    Female: number analyzed (Participants) | 48 | 48 | 96
    Female: 22-29 | 10 | 8 | 18
    Female: 30-39 | 13 | 18 | 31
    Female: 40-49 | 3 | 11 | 14
    Female: 50-59 | 16 | 7 | 23
    Female: 60-70 | 5 | 3 | 8
    Female: <22 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 96
  Male | 48 | 48 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity for male & female participants
  Participants
    Male: number analyzed (Participants) | 48 | 48 | 96
    Male: Hispanic or Latino | 0 | 0 | 0
    Male: Not Hispanic or Latino | 48 | 48 | 96
    Male: Unknown or Not Reported | 0 | 0 | 0
    Female: number analyzed (Participants) | 48 | 48 | 96
    Female: Hispanic or Latino | 0 | 0 | 0
    Female: Not Hispanic or Latino | 48 | 48 | 96
    Female: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Data are presented for both male and female participants
  Participants
    United States | 8 | 10 | 18
    Poland | 52 | 56 | 108
    Georgia | 32 | 28 | 60
    Bulgaria | 4 | 2 | 6
Height [Mean (Standard Deviation); unit: cm] — Population: Data are presented for male participants only as not measured in the females
  cm
    number analyzed (Participants) | 48 | 48 | 96
    (all) | 179.20 (7.24) | 179.43 (7.66) | 179.31 (7.41)
Height [Median (Full Range); unit: cm] — Population: Data are presented for male participants only as not collected in females
  cm
    number analyzed (Participants) | 48 | 48 | 96
    (all) | 177.50 [167.0 to 196.0] | 180.00 [156.0 to 194.0] | 179.00 [156.0 to 196.0]
Weight [Mean (Standard Deviation); unit: kg] — Population: Data are presented for male participants only and not measured in females
  kg
    number analyzed (Participants) | 48 | 48 | 96
    (all) | 88.84 (15.36) | 88.19 (13.72) | 88.52 (14.49)
Weight [Median (Full Range); unit: kg] — Population: Data are presented for male participants only as not collected for females
  kg
    number analyzed (Participants) | 48 | 48 | 96
    (all) | 85.70 [61.0 to 129.0] | 85.15 [66.2 to 130.0] | 85.35 [61.0 to 130.0]
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Population: Data are presented for male participants only as not determined in females
  kg/m2
    number analyzed (Participants) | 48 | 48 | 96
    (all) | 27.643 (4.348) | 27.459 (4.372) | 27.551 (4.338)
Body Mass Index [Median (Full Range); unit: kg/m2] — Population: Data are presented for male participants only as not determined in females
  kg/m2
    number analyzed (Participants) | 48 | 48 | 96
    (all) | 26.985 [18.62 to 39.64] | 26.759 [19.30 to 43.12] | 26.959 [18.62 to 43.12]
Baseline Erectile Dysfunction (ED) severity [Count of Participants; unit: Participants] — Mild ED = IIEF-EF domain score of 17-25, Moderate ED = IIEF-EF domain score of 11-16, Severe ED = IIEF-EF domain score of <= 10. Population: Data are presented for male participants only as not relevant for females
  Participants
    number analyzed (Participants) | 48 | 48 | 96
    Mild | 19 | 19 | 38
    Moderate | 17 | 17 | 34
    Severe | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Erectile Function (EF) Domain of the International Index of Erectile Function (IIEF) Questionnaire, in Patients Randomised to MED3000, at Week 24
Description: Co-primary objectives:
  * Demonstrate an improvement compared to baseline of erectile function, in patients randomised to receive MED3000, using the IIEF-EF patient reported outcome instrument.
  * Observe a mean change from baseline of the IIEF-EF, in patients randomised to MED3000, greater or equal to the minimal clinically importance difference of 4.
  The IIEF is a validated questionnaire, consisting of 15 questions, for detecting treatment changes in EF. The EF domain of IIEF is derived using questions 1, 2, 3, 4, 5 and 15. A score of 0 to 5 is awarded to each of questions 1 to 5 and a score of 1 to 5 is awarded to question 15. Higher scores indicate better sexual function. Domain score is computed by summing the scores for individual questions. The minimum and maximum possible scores are 1 and 30 respectively. Patients with a score of 21 or less are considered to have ED. Change from baseline = Week 24 score - Baseline score.
Time Frame: Baseline and Week 24
Population: MED3000 randomised patients (the only group considered for this outcome). Week 24 values for patients who do not have a Week 24 IIEF-EF value due to early treatment discontinuation adversely related to randomised treatment were imputed as baseline value resulting in zero change from baseline. Week 24 values for patients with early termination discontinuation not adversely related to randomised treatment were imputed via multiple imputation method.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | MED3000
Number analyzed (Participants) | 48
Score on a scale | 5.73 (1.00)
Statistical Analysis 1: Comparison: MED3000; Null hypothesis: mu <= 0 versus alternative hypothesis: mu >0, where mu is the population mean change from baseline in the EF domain of the IIEF questionnaire at week 24; Test type: Other; p < 0.001, t-test, 1 sided — Significance level of 0.025

2. Secondary Outcome: Percentage of Uses Per Patient That Led to an Onset of Erection Within a Certain Period of Time in Patients Randomised to MED3000.
Description: Demonstrate a speed of onset of action from application of MED3000 gel to the time when patient notices their erection starting.
  Percentage of MED3000 uses per patient that resulted in the patient noticing their erection starting within certain period of time, out of the total number of intercourse attempts made using the product during the 24-week treatment period. The certain periods of time are within 15 minutes, 10 minutes and 5 minutes. Percentage of uses is calculated with the denominator equal to the total number of intercourse attempts made using the product during the 24-week treatment period and the numerator equal to the total number of times that the response to the onset of action question 1 indicated a time of 5 (10, 15) minutes or less.
  Question 1 of the Onset of Action questionnaire:
  - After application of the gel/taking medication, when did you begin to notice your erection starting?
Time Frame: 24 weeks
Population: MED3000 randomised patients (the only group considered for this outcome)
Measure: Mean (Standard Deviation); unit: percentage of uses per patient
Arm/Group | MED3000
Number analyzed (Participants) | 48
percentage of uses per patient
  15 minutes | 62.59 (39.18)
  10 minutes | 47.81 (36.26)
  5 minutes | 24.01 (33.43)
Statistical Analysis 1: Comparison: MED3000; Null hypothesis: mu <= 30 versus alternative hypothesis: mu >30, where mu is the population mean percentage of MED3000 uses per patient that resulted in the patient noticing their erection starting within 15 minutes; Test type: Other; p < 0.001, t-test, 1 sided — Significance level of 0.025
Statistical Analysis 2: Comparison: MED3000; Null hypothesis: mu <= 30 versus alternative hypothesis: mu >30, where mu is the population mean percentage of MED3000 uses per patient that resulted in the patient noticing their erection starting within 10 minutes; Test type: Other; p < 0.001, t-test, 1 sided — Significance level of 0.025
Statistical Analysis 3: Comparison: MED3000; Null hypothesis: mu <= 30 versus alternative hypothesis: mu >30, where mu is the population mean percentage of MED3000 uses per patient that resulted in the patient noticing their erection starting within 5 minutes; Test type: Other; p = 0.890, t-test, 1 sided — Significance level of 0.025

3. Secondary Outcome: Percentage of Uses Per Patient That Led to an Onset of Action Within a Certain Period of Time in Patients Randomised to MED3000.
Description: Demonstrate a speed of onset of action from application of MED3000 gel to the time when the patients is able to have penetrative sex.
  Percentage of MED3000 uses per patient that resulted in the patient being able to have penetrative sex within certain period of time, out of the total number of intercourse attempts made using the product during the 24-week treatment period. The certain periods of time are within 15 minutes, 10 minutes and 5 minutes. Percentage of uses is calculated with the denominator equal to the total number of intercourse attempts made using the product during the 24-week treatment period and the numerator equal to the total number of times that the response to the onset of action question 2 indicated a time of 5 (10, 15) minutes or less.
  Question 2 of the Onset of Action questionnaire:
  - After application of the gel/taking medication, when were you able to have penetrative sex?
Time Frame: 24 weeks
Population: MED3000 randomised patients (the only group considered for this outcome)
Measure: Mean (Standard Deviation); unit: percentage of uses per patient
Arm/Group | MED3000
Number analyzed (Participants) | 48
percentage of uses per patient
  15 minutes | 55.70 (36.13)
  10 minutes | 31.91 (29.30)
  5 minutes | 13.72 (22.33)
Statistical Analysis 1: Comparison: MED3000; Test type: Other; p < 0.001, t-test, 1 sided — Significance level of 0.025
Statistical Analysis 2: Comparison: MED3000; Test type: Other; p = 0.3327, t-test, 1 sided — Significance level of 0.025
Statistical Analysis 3: Comparison: MED3000; Test type: Other; p > 0.999, t-test, 1 sided — Significance level of 0.025

ADVERSE EVENTS:
Time Frame: 29 Weeks
Description: Both patients and their female partners were monitored for AEs in the study. In the Other (not including SAE) section, AEs have been separated into those experienced by males and those experienced by their females. For this reason the risk value is recorded as 47 in this section. However, the risk value in the SAE and All-mortality sections is 94 which represents both the male and female participants combined.
Arm/Group | MED3000 | Tadalafil
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94 | 1/94
Other Adverse Events (participants affected / at risk) | 10/47 | 16/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MED3000 (N=94) | Tadalafil (N=94)
Appendicitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MED3000 (N=47) | Tadalafil (N=47)
Nausea (Male) (Gastrointestinal disorders) | 2 | 0
Non-cardiac chest pain (Male) (General disorders) | 0 | 2
Back Pain (Male) (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Male) (Nervous system disorders) | 2 | 9
Headache (Female) (Nervous system disorders) | 3 | 0
Abdominal distension (Male) (Gastrointestinal disorders) | 1 | 1
Gamma-glutamyltransferase increased (Male) (Investigations) | 1 | 1
Pain in extremity (Male) (Musculoskeletal and connective tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion, the results of the clinical investigation (CI) may be published (first publication shall be referred to as the "Primary Paper"). Results of the CI shall not be published before the primary paper after which PIs may propose publications, including or based on results of the CI, to the Sponsor for review at least 2 months before the planned submission for publication or public disclosure. The Sponsor will provide written approval or reasoned refusal for submission or disclosure.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04984993/Prot_SAP_002.pdf